CLINICAL TRIAL: NCT02321982
Title: Same-day Versus Separate-day Preoperative Consultation for Mohs Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study topic is no longer being pursued by study team members
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: D15025
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Non-melanoma Skin Cancer; Squamous Cell Carcinoma of Skin; Basal Cell Carcinoma
Keywords: Mohs surgery; Preoperative consultation
MeSH Terms: conditions — Carcinoma, Basal Cell

ARMS (2):
- Separate-day preoperative consultation (No Intervention): Patients referred for Mohs surgery for non-melanoma skin cancer will have a preoperative consultation in advance of the day of the procedure.
- Same-day preoperative consultation (Experimental): Patients referred for Mohs surgery for non-melanoma skin cancer will have a preoperative consultation on the day same day as the procedure.
  Interventions: Other: Same-day preoperative consultation

INTERVENTIONS:
Other: Same-day preoperative consultation — Preoperative consultation occurs on the same day as Mohs surgery
  Arms: Same-day preoperative consultation

SUMMARY:
The purpose of this study is to determine whether separate- versus same-day preoperative consultation affects time to treatment (start to finish), utilization rate of Mohs, rate of case cancellations, cost, and patient satisfaction. The investigators hypothesize that patients with same-day preoperative consultation will have a shorter time between cancer diagnosis and removal but, only when coordination of care is needed, longer time between removal and consultation with other specialists, as compared to patients with separate-day consultation. The investigators anticipate that patients with same-day preoperative consultation will have a decrease in travel cost as compared to patients with separate-day consultation. The investigators expect that there will be no difference in various satisfaction matters between groups, with the exception of potentially greater convenience reported by patients in the same-day preoperative consultation group. Finally, the investigators hypothesize that there will be no difference between groups in regards to rates of surgery cancellation.

DETAILED DESCRIPTION:
Procedure: Prospective trial which randomly assigns patients to either separate- or same-day preoperative consultation for Mohs surgery. A phone consultation will take place, which will assist in determining whether the patient is appropriate for enrollment into the study. If so, the patient will be randomized to either separate-day or same-day preoperative consultation.

Materials: Patient survey

Methods of data collection: The patient-specific data obtained from the medical record will include: Patient age, number of previous skin cancers, preoperative size, history of cutaneous surgery, employment status, and distance between home address and dermatology facility. Outcome measures that will be obtained from the medical record will include: Time between cancer diagnosis, removal and defect repair, rate of proceeding with Mohs as opposed to other treatment options, and rate of cancelling surgery (due to site discrepancy, anticoagulation issues). A survey will be used to assess patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be considered for enrollment if they have been referred to a Mohs surgeon for consideration of Mohs surgery for non-melanoma skin cancer

Exclusion Criteria:

* Patients would be excluded if there is a lack of indication for Mohs
* Significant comorbidities, or
* In the case of a high-risk location or tumor size, for which in advance it is known that they will need consultation with other specialties

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
Time to treatment | Eight weeks
  Assess the total amount of time elapsed between skin cancer diagnosis and defect repair
Time to consultation with other specialties | Eight weeks
  Assess the amount of time between cancer diagnosis and consultation with non-dermatologic specialties
Time to repair | Eight weeks
  Assess the amount of time elapsed between cancer removal and defect repair
Patient satisfaction | Eight weeks
  Administer a survey to assess patient's perception of convenience, level of comfort with the procedure, and self-evaluation of knowledge regarding the diagnosis and treatment

SECONDARY OUTCOMES:
Utilization rate of Mohs surgery | Eight weeks
  Assess the percentage of patients who actually proceed with undergoing Mohs surgery in each arm
Rate of case cancellation | Eight weeks
  Assess the number of cases that are cancelled due to site discrepancy, anticoagulation or other medical issues in each arm
Travel cost | Eight weeks
  Assess the total distance traveled by each patient coming and going to Mohs appointment(s)

CONTACTS AND LOCATIONS:
Overall Officials: Faramarz Samie, MD, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center